CLINICAL TRIAL: NCT05803863
Title: Efficacy Comparison of 2 Low-dose Atropine Eye Drops in Vietnamese Children Myopia Management
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Thi Mong Dung Nguyen, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 137221050
Record Dates: First submitted 2023-03-25; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Myopia
Keywords: myopia control; low-dose atropin; Vietnamese children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myatro (Experimental): Prescribing one 0,01% Myatro (Atropine) drop/eye/night , in 12 months Then wash-out in next 12 months
  Interventions: Drug: Myatro
- Myatro XL (Experimental): Prescribing one 0,05% Myatro XL (Atropine) drop/eye/night , in 12 months Then wash-out in next 12 months
  Interventions: Drug: Myatro XL
- Conventional spectacles (No Intervention): Prescribing conventional spectacles and follow-up in 24 months.

INTERVENTIONS:
Drug: Myatro — myopia control with 0.01% atropine drops
  Other Names: Atropine 0.01%
  Arms: Myatro
Drug: Myatro XL — myopia control with 0.05% atropine drops
  Other Names: Atropine 0.05%
  Arms: Myatro XL

SUMMARY:
The goal of this clinical trial is to compare the efficacy of 2 low-dose atropine drops (0,01%; 0,05%) in Vietnamese children. The main questions it aims to answer are:

1. How is the difference in efficacy among 3 groups: atropine 0,01% vs 0,05% vs spectacles?
2. How is the difference in side effects among 3 groups: atropine 0,01% vs 0,05% vs spectacles?
3. How is the difference in rebound phenomena between 2 atropine groups?

DETAILED DESCRIPTION:
The study is prospective, comparative, open label. Participants are Vietnamese children. Prescribing drops : 1 drops/eye/night/ 12 months Wash-out: 12 months The atropine drops in this study are commercially available.

ELIGIBILITY:
Inclusion Criteria:

* myopic 2 eyes (SE above from -0.75 D, astigmatism below -1.50D)
* 8 - 13 years old
* Vietnamese, speaking Vietnamese
* BCVA from 8/10 each eye

Exclusion Criteria:

* Using any contact lens in less than 3 months
* Other eye diseases than myopia
* History of eye trauma, surgeries
* Having chronic systemic diseases or having medications affecting eye.
* Having contraindications of atropine drops
* Pre-known allergies to atropine drops
* Undergoing another myopia control treatments

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy (SE) of Atropine drops | 12 months
  measured by change in spherical equivalent (D) (Objective cycloplegic refraction)
Efficacy (AL) of Atropine drops | 12 months
  axial length (mm)

SECONDARY OUTCOMES:
pupil size | 12 months
  change in pupil size (mm)
amplitude of accommodation | 12 months
  change in amplitude of accommodation (D)
adverse symptoms 1 | 12 months
  rate of photophobia
adverse symptoms 2 | 12 months
  rate of reading difficulties
rebound effect (SE) | 12 months
  change in spherical equivalent (D) after wash-out (Objective cycloplegic refraction)
rebound effect (AL) | 12 months
  change in axial length(mm) after wash-out

CONTACTS AND LOCATIONS:
Overall Officials: Dung TM Nguyen, MD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University Medical Center HCMC, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No